CLINICAL TRIAL: NCT06425991
Title: A Phase 1 Randomized, Open Label Pharmacokinetic Comparability Study Comparing Pre- and Post-change Teclistamab in Participants With Relapsed/Refractory Multiple Myeloma
Brief Title: A Study Comparing Pre- and Post-Change Teclistamab in Participants With Relapsed or Refractory Multiple Myeloma
Acronym: MajesTEC-10
Status: Active, not recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Janssen Research & Development, LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 64007957MMY1008; 64007957MMY1008 (Other: Janssen Research & Development, LLC); 2023-508426-10-00 (Registry Identifier: EUCT number)
Record Dates: First submitted 2024-05-17; First posted 2024-05-23 (Actual); Last update posted 2026-01-16 (Actual); Status verified 2026-01

CONDITIONS: Relapsed or Refractory Multiple Myeloma
Keywords: 1-3 prior lines
MeSH Terms: conditions — Recurrence; Multiple Myeloma

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Arm A: Pre-change Teclistamab (Experimental): Participants will receive teclistamab monotherapy (made from the pre-change manufacturing process) for all step-up and treatment doses until confirmed progressive disease, death, intolerable toxicity, withdrawal of consent to treatment, or end of the study, whichever occurs first.
  Interventions: Drug: Teclistamab
- Arm B: Post-change Teclistamab (Experimental): Participants will receive teclistamab monotherapy (made from the post-change manufacturing process) for all step-up and treatment doses until confirmed progressive disease, death, intolerable toxicity, withdrawal of consent to treatment, or end of the study, whichever occurs first.
  Interventions: Drug: Teclistamab

INTERVENTIONS:
Drug: Teclistamab — Teclistamab will be administered subcutaneously.
  Other Names: JNJ-64007957

SUMMARY:
The purpose of this study is to compare the pharmacokinetics (processes by which drugs are absorbed, distributed in the body, and excreted) between teclistamab made from the current commercial manufacturing process (pre-change) and the new manufacturing process (post-change).

ELIGIBILITY:
Inclusion Criteria:

* Documented diagnosis of multiple myeloma as defined by the criteria below: (a) Multiple myeloma diagnosis according to International Myeloma Working Group (IMWG) diagnostic criteria (b) Measurable disease at screening as defined by any of the following: (1) Serum M-protein level greater than or equal to (>=) 0.5 grams per deciliter (g/dL) (central laboratory); or (2) Urine M-protein level >=200 milligrams (mg)/24 hours (central laboratory); or (3) Serum immunoglobulin free light chain >=10 milligrams per deciliter (mg/dL) (central laboratory) and abnormal serum immunoglobulin kappa lambda free light chain ratio
* Received 1 to 3 prior lines of antimyeloma therapy, including a minimum of 2 consecutive cycles each of a protease inhibitor (PI), lenalidomide, and an anti-cluster of differentiation 38 (CD38) monoclonal antibody (or minimum of 6 doses if anti CD38 monoclonal antibody was only part of a maintenance regimen) in any prior line
* Documented evidence of progressive disease or failure to achieve a response to last line of therapy based on investigator's determination of response by IMWG criteria
* Have an eastern cooperative oncology group (ECOG) performance status score of 0 to 2
* A female participant of childbearing potential must have a negative highly sensitive serum pregnancy test at screening and within 24 hours of the start of study treatment and must agree to further serum or urine pregnancy tests during the study

Exclusion Criteria:

* Received any bispecific antibody and/or chimeric antigen receptor T cell (CAR-T) cell therapy
* Contraindications or life-threatening allergies, hypersensitivity, or intolerance to any study drug or its excipients
* Received a live, attenuated vaccine within 4 weeks before the first dose of study drug. Non-live or non-replicating vaccines authorized for emergency use by local health authorities are allowed
* Central nervous system involvement or clinical signs of meningeal involvement of multiple myeloma. If either is suspected, negative whole brain magnetic resonance imaging (MRI) and lumbar cytology may be required
* Participant had major surgery or had significant traumatic injury within 2 weeks prior to randomization, or will not have fully recovered from surgery, or has major surgery planned during the time the participant is expected to be treated in the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 108 (Actual)
Dates: Start 2024-06-07 (Actual); Primary Completion 2027-02-28 (Estimated); Study Completion 2027-03-03 (Estimated)

PRIMARY OUTCOMES:
Maximum Observed Serum Concentration (Cmax) of First Treatment Dose of Teclistamab | Cycle 1 (28 days cycle): Predose to Day 7 postdose
  Cmax is defined as the maximum observed serum concentration of teclistamab (after first treatment dose).
Area Under Serum Concentration Versus Time Curve (AUCtau) of Teclistamab First Treatment Dose | Cycle 1 (28 days cycle): Predose to Day 7 postdose
  AUCtau is defined as area under the concentration-time curve during dosing interval of teclistamab (after first treatment dose).
Observed Serum Concentration Immediately Prior to the Next Study Treatment Administration (Ctrough) on Cycle 3 Day 1 | Cycle 3 (28 days cycle): Day 1
  Ctrough is defined as observed serum concentration immediately prior to the next study treatment administration.

SECONDARY OUTCOMES:
Number of Participants with Anti-drug Antibodies (ADAs) | Up to approximately 3 years
  Number of participants with ADAs to teclistamab will be reported.
Percentage of Participants With Complete Response (CR) or Better Response | Up to approximately 3 years
  Percentage of participants with CR or better response will be reported. CR or better response rate is defined as participants who achieve a CR or better response prior to subsequent antimyeloma therapy in accordance with the IMWG criteria.
Number of Participants with Adverse Events (AEs) by Severity | Up to approximately 3 years
  An adverse event is any untoward medical occurrence in a clinical study participant administered a pharmaceutical (investigational or non-investigational) product. An adverse event does not necessarily have a causal relationship with the treatment. Severity will be graded according to the National Cancer Institute Common Terminology Criteria for Adverse Events (NCI-CTCAE) version 5.0. Severity scale ranges from Grade 1: mild, Grade 2: moderate, Grade 3: severe, Grade 4: life-threatening, and Grade 5: death related to adverse event.
Number of Participants with Serious Adverse Events (SAEs) | Up to approximately 3 years
  SAEs are any AE which results in death, is life-threatening, requires inpatient hospitalization or prolongation of existing hospitalization, results in persistent or significant disability/incapacity, is a congenital anomaly/birth defect, is a suspected transmission of any infectious agent via a medicinal product, or is medically important.
Number of Participants with Abnormal Laboratory Results | Up to approximately 3 years
  Number of participants with abnormal laboratory results (such as hematology and chemistry) will be reported.
Percentage of Participants With Overall Response (Partial Response [PR] or Better) | Up to approximately 3 years
  Percentage of participants with overall response (PR or better) will be reported. Overall response (PR or better) is defined as participants who have a PR or better prior to subsequent antimyeloma therapy in accordance with the international myeloma working group (IMWG) criteria.
Percentage of Participants With Very Good Partial Response (VGPR) or Better Response | Up to approximately 3 years
  Percentage of participants with VGPR or better response will be reported. VGPR or better response rate is defined as participants who achieve a VGPR or better response prior to subsequent antimyeloma therapy in accordance with the IMWG criteria.

CONTACTS AND LOCATIONS:
Overall Officials: Janssen Research & Development, LLC Clinical Trial, Study Director — Janssen Research & Development, LLC
Locations (53):
- United States (7):
  - Banner MD Anderson Cancer Center, Gilbert, Arizona
  - Colorado Blood Cancer Institute, Denver, Colorado
  - Cleveland Clinic Florida, Weston, Florida
  - Augusta University- Georgia Cancer Center, Augusta, Georgia
  - St Francis Hospital & Health Centers Indiana Blood and Marrow Transplantation Franciscan Health, Indianapolis, Indiana
  - Cleveland Clinic, Cleveland, Ohio
  - Baylor University Medical Center, Dallas, Texas
- Australia (4):
  - Flinders Medical Centre, Bedford Park
  - Box Hill Hospital, Box Hill
  - Royal Prince Alfred Hospital, Camperdown
  - Epworth Healthcare, Richmond
- Canada (2):
  - Cross Cancer Institute, Edmonton, Alberta
  - Princess Margaret Cancer Centre University Health Network, Toronto, Ontario
- France (4):
  - CHRU de Lille Hopital Claude Huriez, Lille
  - CHU Nantes, Nantes
  - CHU de Bordeaux - Hospital Haut-Leveque, Pessac
  - CHU Lyon Sud, Pierre-Bénite
- Germany (4):
  - Klinikum Chemnitz gGmbH, Chemnitz
  - Universitaetsklinikum Hamburg Eppendorf, Hamburg
  - Universitaetsklinikum Heidelberg, Heidelberg
  - Universitatsklinikum Wurzburg, Würzburg
- Israel (4):
  - Carmel Medical Center, Haifa
  - Hadassah University Hospita Ein Kerem, Jerusalem
  - Sheba Medical Center, Ramat Gan
  - Sourasky Medical Center, Tel Aviv
- Italy (6):
  - Ospedali Riuniti Di Ancona, Ancona
  - ASST Papa Giovanni XXIII Bergamo, Bergamo
  - Azienda Ospedaliera Spedali Civili di Brescia, Brescia
  - Istituto Scientifico Romagnolo per lo Studio e la Cura dei Tumori, Meldola
  - Ospedale Santa Chiara AO Universitaria Pisana, Pisa
  - Policlinico Universitario Agostino Gemelli, Rome
- Poland (6):
  - Wojewodzki Szpital Specjalistyczny, Biała Podlaska
  - Uniwersyteckie Centrum Kliniczne, Gdansk
  - Pratia Onkologia Katowice, Katowice
  - Swietokrzyskie Centrum Onkologii SPZOZ w Kielcach, Kielce
  - Centrum Onkologii Ziemi Lubelskiej im sw Jana z Dukli, Lublin
  - Dolnoslaskie Centrum Onkologii, Wroclaw
- South Korea (5):
  - Seoul National University Hospital, Seoul
  - Severance Hospital Yonsei University Health System, Seoul
  - Asan Medical Center, Seoul
  - Samsung Medical Center, Seoul
  - The Catholic University of Korea Seoul St Mary s Hospital, Seoul
- Spain (7):
  - Hosp Clinic de Barcelona, Barcelona
  - ICO L'Hospitalet - Hospital Duran i Reynals, Barcelona
  - Hosp. Univ. 12 de Octubre, Madrid
  - Clinica Univ. de Navarra, Pamplona
  - Hosp. Quiron Madrid Pozuelo, Pozuelo de Alarcón
  - Hosp Clinico Univ de Salamanca, Salamanca
  - Hosp. Univ. Marques de Valdecilla, Santander
- United Kingdom (4):
  - Hammersmith Hospital, London
  - The Christie NHS Foundation Trust Christie Hospital, Manchester
  - Norfolk & Norwich University Hospital, Norwich
  - Derriford Hospital, Plymouth

IPD SHARING:
Plan to Share IPD: Yes
The data sharing policy of the Janssen Pharmaceutical Companies of Johnson & Johnson is available at www.janssen.com/clinical-trials/transparency. As noted on this site, requests for access to the study data can be submitted through Yale Open Data Access (YODA) Project site at yoda.yale.edu
URL: https://www.janssen.com/clinical-trials/transparency